CLINICAL TRIAL: NCT05188456
Title: The Impact Evaluation of the COVID-19 Prevention Knowledge, Attitude, and Practice on Risk Factors of HIV and Sexually Transmitted Comorbidity: Application of Protection Motivation Theory
Brief Title: The Impact Evaluation of the COVID-19 Prevention on Risk Factors of HIV and Sexually Transmitted Comorbidity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Other Study IDs: 202012HM041
Record Dates: First submitted 2022-01-10; First posted 2022-01-12 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pandemics; Human Immunodeficiency Virus
Keywords: Attitude; Behavior; Coronavirus disease 19 (COVID-19); HIV high risk group; Knowledge; People living with HIV/AIDS (PLWHA); Protection Motivation Theory (PMT); Stigma
MeSH Terms: conditions — COVID-19; Acquired Immunodeficiency Syndrome; Behavior; Social Stigma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional research. The Protection Motivation Theory (PMT) was applied as theoretical framework to analyze correlation of prevention knowledge, prevention intentions and anxiety, and prevention behavior of COVID-19 and HIV risk feature and behavior and stigma of people living with HIV/AIDS (PLWHA), and HIV high-risk groups. Purposive and snowball sampling will be applied to recruit participant who visit hospital, HIV/AIDS related institutions, and social media platforms. The investigators expect that the outcome could reveal the relationship of cognition and attitude of COVID-19 to HIV prevention and treatment.

DETAILED DESCRIPTION:
The prevention strategies can effectively block the spread of Coronavirus disease (Coronavirus disease 19; COVID-19), and at the same time may indirectly reduce or increase the risk behaviors and factors of Human Immunodeficiency Virus (HIV) and sexually transmitted comorbidities. The main purpose of this research is to apply the Protection Motivation Theory (PMT) as the framework to analyze COVID-19 prevention knowledge, COVID-19 prevention intentions and anxiety level, and COVID-19 prevention behavior and HIV risk behavior and risk factors of people living with HIV/AIDS (PLWHA) and HIV high-risk groups. The cross-sectional research method was adopted, and the subjects included the northern, central, southern, and eastern regions of Taiwan.About 1100 PLWHA and 1100 high-risk groups will be recruited. The information of recruitment will be disseminated through the AIDS designated medical institutions and related institutions, and social media, Snowball recruitment of interviewees will also be used. After completing the online questionnaire, the structural equation modeling (SEM) will be applied to test the good of fit of the theory model and to explain the structural relationship between COVID-19 prevention knowledge, attitudes, behaviors and HIV risk factors. The relationship with the above variables and stigma also been discussed. In addition to verifying the theories proposition of PMT, the research results also contribute to the prevention and treatment of HIV high-risk groups, and provide important references for prevention strategies for susceptible groups during the epidemic of emerging infectious diseases in the future.

ELIGIBILITY:
Inclusion Criteria for HIV/AIDS participants:

1. Participants who diagnosed with HIV/AIDS.
2. Age over 18 years old.
3. Participants who can read and communicate.

Exclusion Criteria for HIV/AIDS participants:

1. Participants who can't read and communicate.

Inclusion Criteria for HIV high risk group:

1. Participants who have experienced unsafe sex, regardless of their gender orientation, such as those who describe themselves as men who have sex with men (MSM), heterosexuals, transgender, sex workers, etc.
2. Injecting Drug User(IDU)
3. Age over 18 years old.
4. Participants who can read and communicate.

Exclusion Criteria for HIV high risk group:

1. Participants who can't read and communicate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two study populations will be incruited in this research:
  1. Those who had been diagnosed with HIV/AIDS.
  2. Those who self-idenftified as HIV high risk group, such as having unsafe sex experience or injecting drug user.
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 prevention knowledge | Through study completion, an average of one and half year
  The questionnaire of COVID-19 prevention knowledge will be used to measure the knowledge level.
COVID-19 prevention intention and anxiety | Through study completion, an average of one and half year
  The questionnaire of COVID-19 prevention intention and anxiety will be used to measure the attitude level.
COVID-19 prevention behavior | Through study completion, an average of one and half year
  The questionnaire of COVID-19 prevention behavior will be used to measure the behavior level.
Stigma | Through study completion, an average of one and half year
  The questionnaire of stigma will be used to measure the stigma level of HIV infected people.
HIV risk factor and behavior | Through study completion, an average of one and half year
  The questionnaire of HIV risk factor and behavior will be used to measure the risk condition during COVID-19 era.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing of National Taiwan University, Taipei, Taiwan